CLINICAL TRIAL: NCT04181710
Title: Evaluation of a Marine OXYgen Carrier for Organ Preservation : a Multicenter Randomized Study Evaluating the Efficacy of HEMO2life® Versus Standard of Care in Renal Transplantation
Brief Title: Evaluation of a Marine OXYgen Carrier for Organ Preservation
Acronym: OXYOP 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OXYOP 2 (29BRC19.0048)
Record Dates: First submitted 2019-11-27; First posted 2019-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: End Stage Renal Diseases
Keywords: Kidney transplantation; Organ preservation
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEMO2life (Experimental): HEMO2life® will be used for ex vivo graft preservation at the dose of 1g per liter of preservation solution.
  Interventions: Procedure: Kidney transplant
- Control (Other): Organ preserved in preservation solution routinely used according to the local practice
  Interventions: Procedure: Kidney transplant

INTERVENTIONS:
Procedure: Kidney transplant — Organ preserved in preservation solution

SUMMARY:
Preventing ischemia/reperfusion injuries (IRIs) is a major issue in kidney transplantation, particularly for transplant recipients receiving a kidney from extended criteria donors (ECD). The main consequence of IRIs is delayed graft function (DGF).

The medical device HEMO2life®, an oxygen carrier developed by the Hemarina French Company, is a natural extracellular hemoglobin (Hb) isolated from the marine lugworm Arenicola marina. This biopolymer of high molecular weight (~3,600 kDa) has a large oxygen binding capacity, carrying up to 156 oxygen molecules when saturated (4 for human Hb). It releases oxygen according to a simple gradient and exhibits an intrinsic superoxide dismutase-like activity preventing both the occurrence of potentially harmful heme-protein-associated free radical species and the release of Hb degradation products.

Recently a safety study in 60 renal grafts using HEMO2life® as additive to organ preservation solution (Oxyop study, NCT02652520) was completed, that confirmed that the use of HEMO2life® is safe for patients and grafts.

In the Oxyop study, even if the protocol was not designed to show a benefit of the use of HEMO2life®, significantly less delayed graft function (DGF) and a shorter renal function recovery was observed.

The present research focuses on the efficacy of HEMO2life®, which is an oxygen carrier added in preservation solution in kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* For Kidney graft:
* Any pair of kidneys retrieved in an adult donor in one of first line participating centers.
* Any pair of kidneys from a deceased donor after brain or cardiac death
* For Patient:
* Male or female renal allograft recipients at least 18 years old
* Patient who signed an inform consent form
* Patient receiving one graft from an included pair of kidneys

Exclusion criteria :

* For kidney :
* Graft from a living donor
* Graft dedicated to a multi-organ transplantation or dual kidney transplantation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of HEMO2life® as an additive to standard organ preservation solution to prevent delayed graft function following renal transplantation. | From day 0 to day 7
  Delayed graft function defined as the requirement for dialysis during the first week after transplantation will be compared as per the confirmatory testing strategy

SECONDARY OUTCOMES:
Assess and compare graft and patient survival in the two groups. | From month 0 to month 12
  Graft and patient survival at one year
Efficacy of HEMO2life® on renal parameters compared with standard of care | From month 0 to month 12
  Evaluation using DGF assessed with alternative definitions: more than one dialysis session, need for dialysis except for hyperkaliemia or overhydration reason, time to reach a creatinine value of 250 µmol/l, DGF duration and using Renal function (creatinine value and eGFR)
Efficacy in specific populations depending on type of donors and the type of preservation solution. | From month 0 to month 12
  Rate of primary non function
Evaluate the impact of HEMO2Life® on the degree and progression of interstitial fibrosis on the pre-implantation and 3 month biopsies | biopsies pre-implantation and month 3
  Rate of biopsy-proven acute rejection at one year
Evaluate the impact of HEMO2life® on quality of life following renal transplant at Month-1, 3 and 12. | From Day 0 to month 12
  Quality of life assess using the generic self-administered questionnaire EuroQol-5 Dimensions (EQ-5D) and a specific questionnaire for renal transplant recipients in the French language: the ReTransQol (RTQ) [0-100]. For RTQ, higher score mean a better outcome.
Safety profile of HEMO2life® post transplant | From organ preservation to month 12
  Safety profile of HEMO2life® post transplant based on 3 analysis : graft safety, recipient safety, graft function

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MEUR, Principal Investigator — Principal Investigator and Nephrology coordinator; Benoit BARROU, Principal Investigator — Urology coordinator
Locations (32):
- France (32):
  - Amiens, Amiens
  - Angers, Angers
  - Besançon, Besançon
  - Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - Caen, Caen
  - Clermont-Ferrand, Clermont-Ferrand
  - Dijon, Dijon
  - Grenoble, Grenoble
  - Lille, Lille
  - Limoges, Limoges
  - Lyon, Lyon
  - Marseille, Marseille
  - Montpellier, Montpellier
  - Nancy, Nancy
  - Nantes, Nantes
  - Nice, Nice
  - APHP Bicêtre, Paris
  - APHP Henri Mondor, Paris
  - APHP Necker, Paris
  - APHP Saint-Louis, Paris
  - Association Hopital Foch, Paris
  - Paris La Salpétrière, Paris
  - Poitiers, Poitiers
  - Reims, Reims
  - Rennes, Rennes
  - Rouen, Rouen
  - La Réunion, Saint-Denis
  - Saint-Etienne, Saint-Etienne
  - Strasbourg, Strasbourg
  - Toulouse, Toulouse
  - Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743
- [Derived] Le Meur Y, Nowak E, Barrou B, Thierry A, Badet L, Buchler M, Rerolle JP, Golbin L, Duveau A, Dantal J, Merville P, Kamar N, Demini L, Zal F. Evaluation of the efficacy of HEMO2life(R), a marine OXYgen carrier for Organ Preservation (OxyOp2) in renal transplantation: study protocol for a multicenter randomized trial. Trials. 2023 May 1;24(1):302. doi: 10.1186/s13063-023-07302-3. PMID 37127632